CLINICAL TRIAL: NCT03167697
Title: Evaluating the Efficacy of PKU Synergy in Patients Expressing Phenylketonuria or Hyperphenylalaninemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PKUSyn.2017
Record Dates: First submitted 2017-05-22; First posted 2017-05-30 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Phenylketonurias; Hyperphenylalaninaemia, Type I
Keywords: Phenylketonuria; Hyperphenylalaninaemia; Inherited Metabolic Disorders
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synergy (Experimental): This group will receive the new phenylalanine-free protein substitute daily for 28 days. Patients in this group intervention will be directed to consume one powder sachet (33 g) of daily made up with 100mL of water. The new substitute delivers 414 kJ, 20g protein equivalent and a combination of essential and non-essential amino acids as well a combination of vitamins and minerals.
  Interventions: Dietary Supplement: Synergy
- Routine (Active Comparator): This group will continue their usual dietary and/or protein substitute regimen (maximum of 1 protein substitute per day (equal to 20g protein equivalent) control) for 28 days.
  Interventions: Other: Routine

INTERVENTIONS:
Dietary Supplement: Synergy — Small serving (x1 33 g serving daily) of the new phenylalanine-free protein substitute made up with 100mL of water daily (28 days).
  Arms: Synergy
Other: Routine — Patients will continue their usual dietary and/or protein substitute regimen (28 days).
  Arms: Routine

SUMMARY:
This study centres around a new one-a-day phenylalanine-free protein substitute for phenylketonuria patients. Fifty eligible adults (≥ 16 years) with proven phenylketonuria or hyperphenylalaninemia will be recruited and randomly allocated to one of two intervention arms (n = 25 per arm). Following a 3-day baseline period, and in addition to routine nutritional management, patients will receive either one sachet of the new protein substitute daily (intervention) or continue their usual dietary and/or protein substitute regimen (maximum of 1 protein substitute per day (equal to 20g protein equivalent) control) for 28 days.

DETAILED DESCRIPTION:
This study centres around a new one-a-day phenylalanine-free protein substitute for phenylketonuria patients. In particular, this randomised controlled trial aims to evaluate the efficacy (changes relating to nutritional status and metabolic control) of this new protein substitute, while also capturing data pertaining to tolerance, compliance, safety and acceptability. Designed for poorly compliant adult patients with proven phenylketonuria or hyperphenylalaninemia, this new protein substitute is composed of an adapted mixture of other essential and non-essential amino acids, carbohydrates, vitamins and selected minerals and trace elements and enriched with docosahexaenoic acid (DHA). Fifty eligible adults (≥ 16 years) will be recruited and randomly allocated to one of two intervention arms (n = 25 per arm). Following a 3-day baseline period, and in addition to routine nutritional management, patients will receive either one sachet of the new protein substitute daily (intervention) or continue their usual dietary and/or protein substitute regimen (maximum of 1 protein substitute per day (equal to 20g protein equivalent) control) for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Over 16 years of age
* Diagnosed with proven PKU or hyperphenylalaninemia with an increased phenylalanine-tolerance/intake
* Currently taking a maximum of 1 protein substitute per day (equal to 20g protein equivalent)
* Have a minimum blood phenylalanine level of ≥ 600 umol/L (for PKU patients)
* Have relaxed (if not stopped) their dietary and protein substitute regimen for at least 1 month prior to trial commencement
* Have Written informed consent from patient

Exclusion Criteria:

* Pregnant or lactating
* Requiring nutritional support (including enteral and parenteral nutrition)
* Major hepatic or renal dysfunction
* Participation in other studies within 1 month prior to entry of this study
* Allergy to any of the study product ingredients, including milk protein or soya
* Investigator concern around willingness/ability of patient to comply with protocol requirements

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Nutritional Status (objective measure) | 2 days
  Blood micro nutrient levels; active Vitamin B12 (holotranscobalamin)

SECONDARY OUTCOMES:
Nutritional Status (Objective measure) | 2 days
  Blood micro nutrient levels; Folate (Folic Acid)
Nutritional Status (Objective measure) | 2 days
  Blood micro nutrient levels; Iron (Ferritin)
Nutritional Status (Objective measure) | 2 days
  Blood micro nutrient levels; Zinc
Nutritional Status (Objective measure) | 2 days
  Blood micro nutrient levels; Vitamin D (25-hydroxyvitamin D)
Nutritional Status (subjective measure) | 6 days
  3 day weighed food diary
Daily compliance with prescribed protein substitute as assessed by standarised questionnaire | 31 days
  Compliance with the recommended intake of the patients previously prescribed protein substitute (during baseline in both groups, and during the study period in the control group) and with the study product during the intervention period will be assessed daily throughout the study. Patients will be asked to record how much of the protein substitute is taken compared to that recommended by their Health Care Professional. The daily amount prescribed by the Health Care Professional managing the patients care will be recorded at the start of the study and any changes to this prescription during the study will be noted. During the intervention period, protein substitute consumption patterns (e.g. timing and amount consumed) will be recorded daily and assessed b y a standardised questionnaire.
Metabolic Control | 2 days
  Blood amino acid levels; Collected samples will be analysed for blood phenylalanine, tyrosine and 16 other proteinogenic amino acids, 2 non-proteinogenic amino acids and 1 amino sulfonic acid.
Gastrointestinal tolerance as assessed by standarised questionnaire | 12 days
  Gastrointestinal tolerance (including diarrhoea, constipation, nausea, vomiting, abdominal pain, bloating, flatulence and burping) will be assessed using a standardised gastrointestinal tolerance questionnaire completed by the patient.
Acceptability as assessed by standarised questionnaire | 2 days
  Acceptability (ease of use and liking) of the patients previously prescribed protein substitute and the study product will be assessed at the end of baseline (day 4) and the end of the intervention period (day 31) using a standardised questionnaire completed by the patient.
Subjective Mood | 3 days
  Profile of mood states questionnaire
Anthropometry | 2 days
  Measures of weight and height will be made during baseline observations (day 1) and at the end of the intervention period (day 31). Weight will be determined to the nearest 0.1 kg, using portable scales shoeless and wearing light weight clothing.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Stratton, PhD, Principal Investigator — Nutricia UK
Locations (6):
- United Kingdom (6):
  - Queen Elizabeth Hospital, Birmingham
  - Royal Hospital for Sick Children, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow
  - Guys & St Thomas' Hospital, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.